CLINICAL TRIAL: NCT02577380
Title: Addressing Gender Based Violence in HIV Testing and Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Population Council # 640
Record Dates: First submitted 2015-10-01; First posted 2015-10-16 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Intimate Partner Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPV/GBV HIV testing and counseling (Experimental): For the randomized controlled trial, first-time antenatal care clients will be randomly assigned to IPV/GBV HTC HIV testing.
  Interventions: Behavioral: IPV/GBV HTC
- Standard HIV testing and counseling (No Intervention): For the randomized controlled trial, first-time antenatal care clients will be randomly assigned to Standard HIV testing and counseling.

INTERVENTIONS:
Behavioral: IPV/GBV HTC — Participants will be interviewed after receiving their services.
  Arms: IPV/GBV HIV testing and counseling

SUMMARY:
The overarching goal of this study is to pilot an approach to HIV testing and counseling (HTC) that addresses intimate partner violence. The results of the study will fill an important gap in the literature and contribute to efforts by Kenyatta National Hospital in Nairobi, Kenya-and the HIV and sexual and reproductive health field globally-to better address intimate partner violence in our work.

ELIGIBILITY:
Inclusion Criteria:

* Lived in the community for at least one year
* Aged 15-49 years
* Satisfy gender requirement

Exclusion Criteria:

* Lack of informed consent

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Comparison of HTC experiences | 10 months
  Number of ANC clients who meet an expected result of a survey with the intervention group (IPV/GBV-HTC) or with the control group (standard HTC). The score is based on answers given to attitudes toward study participant knowledge regarding IPV/GBV; awareness of IPV/GBV services; and agency regarding talking with their partner about HIV testing.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Haberland, MPH, Principal Investigator — Population Council

REFERENCES:
- [Derived] Haberland N, Ndwiga C, McCarthy K, Pulerwitz J, Kosgei R, Mak'anyengo M, Peltz A, Wong VJ, Kalibala S. Addressing Intimate Partner Violence and Power in Intimate Relationships in HIV Testing Services in Nairobi, Kenya. AIDS Behav. 2020 Aug;24(8):2409-2420. doi: 10.1007/s10461-020-02801-9. PMID 32026250